CLINICAL TRIAL: NCT06382246
Title: The Acute Effect of "Exercise Snacks" on Glycemic Responses in Individuals With Type 2 Diabetes: a Randomized Controlled Crossover Trial
Brief Title: The Acute Effect of "Exercise Snacks" on Glycemic Responses in Individuals With Type 2 Diabetes.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H24-Acute-ExSnacks
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized controlled crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (EX): exercise snacks condition (Experimental): Bodyweight-style exercise snacks lasting 1-minute each performed with vigorous effort 4 times per day on two consecutive days.
  Interventions: Other: Exercise snacks
- Control (CON): Non-exercise condition (No Intervention): No structured exercise on two consecutive days.

INTERVENTIONS:
Other: Exercise snacks — Bodyweight-style exercise snacks lasting 1-minute each performed with vigorous effort 4 times per day on two consecutive days.
  Arms: Exercise (EX): exercise snacks condition

SUMMARY:
To conduct a randomized crossover trial to determine the acute impact of exercise snacks on glycemic control in physically inactive individuals living with type 2 diabetes using continuous glucose monitoring.

DETAILED DESCRIPTION:
Participants will perform two, 48-hour experimental conditions separated by 24 hours while wearing a continuous glucose monitor to measure glycemic responses. The order of the trials will be randomized for each participant. The two trials will include an exercise condition (EX) and a control, non-exercise condition (CON). During the EX trial, participants will perform four exercise snacks per day on two consecutive days (i.e., Monday and Tuesday). Each exercise snack will be 1-minute in duration and consist of bodyweight style exercise performed with vigorous effort. During the CON trial, participants will be asked to refrain from any structured exercise during two consecutive days (i.e., Thursday and Friday). All meals will be provided to participants during the two 48-hour trials and will be standardized for a given participant. There will be a one-day wash out period in between the completion of both trials for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-75 years old.
* Have physician-diagnosed type 2 diabetes.
* Currently participating in less than 150 minutes of moderate-to-vigorous intensity aerobic exercise per week.
* Have a body mass index between 18.5 and 40 kg/m2.
* Have had a stable medication dosage and no changes to the number of prescribed medications for at least 6 months.
* Able to maintain current medication doses during the study.
* Able to maintain current physical activity patterns during the study.
* HbA1c is less than or equal to 8.5%.
* Have access to a computer, tablet, or smartphone for intervention delivery and tracking.
* Can travel to McMaster University for in-person laboratory testing visits.
* Can read, write, and understand English.
* Anticipate having access to the internet for the duration of the intervention (i.e., over the next 3-4 months).
* Cleared for exercise participation based on the CSEP Get Active Questionnaire and the Rose Angina Questionnaire.

Exclusion Criteria:

* Taking 4 or more glucose-lowering medications.
* Taking insulin.
* Taking beta-blockers.
* Taking 3 or more commonly prescribed medications for the prevention of cardiovascular disease (e.g., statins, antihypertensives).
* Have had an episode of severe hypoglycemia in the past 6 months (defined as having neurological symptoms consistent with neuroglycopenia and required assistance in treatment by a second party).
* Currently a cigarette smoker.
* Have a chronic musculoskeletal condition that would prevent participation in exercise.
* Have had a recent (within the last 2 years) cardiovascular event that prevents participation in exercise.
* Experience angina upon exertion.
* Have uncontrolled high blood pressure (hypertension) or an atypical blood pressure or pulse rate at rest or during exercise as determined by a physician.
* Have a scheduled surgical procedure within the next 3-4 months that would prevent exercise participation.
* Currently diagnosed with a cardiac or pulmonary disease (e.g., angina, arrythmia, exercise-induced bronchospasm) that would prevent exercise participation.
* Have a psychiatric disorder that could prevent you from completing the study procedures or visits.
* Have donated more than 0.5 L of blood within the last 4 weeks.
* Currently following an extreme diet (e.g., very low carbohydrate/calorie, ketogenic) or taking dietary/nutritional supplements that impact glucose control (e.g., exogenous ketones).
* Currently have diabetic ulcers, peripheral vascular disease, or diabetic neuropathy that will prevent participation in exercise.
* Currently on dialysis.
* Currently participating in another clinical trial that interferes with the study procedures.
* Currently pregnant or planning on becoming pregnant during the intervention (i.e., within the next 3-4 months).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Mean 24-h glucose concentration assessed using continuous glucose monitoring | 48-hour EX trial versus the 48-hour CON trial
  The mean 24-h glucose per trial will be determined as the average of the two 24-h periods during that specific trial.

SECONDARY OUTCOMES:
Time in range determined using continuous glucose monitoring | 48-hour EX trial versus the 48-hour CON trial
  Percentage of time in range (3.9-10 mmol/L)
Time above range determined using continuous glucose monitoring | 48-hour EX trial versus the 48-hour CON trial
  Percentage of time above range (>10 mmol/L)
Time below range determined using continuous glucose monitoring | 48-hour EX trial versus the 48-hour CON trial
  Percentage of time above range (<3.9 mmol/L)
Glycemic variability determined using continuous glucose monitoring | 48-hour EX trial versus the 48-hour CON trial
  Glycemic variability will be assess using the Standard Deviation (SD), mean amplitude of glycemic excursions (MAGE), and the coefficient of variation (CV)
Two-hour glucose area under the curve following standardized breakfast, lunch and dinner meals | 48-hour EX trial versus the 48-hour CON trial
  The incremental area under the curve following breakfast, lunch and dinner (2 h post meal)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No